CLINICAL TRIAL: NCT03492190
Title: Bioavailability of Proteins From Beans Usually Consumed in the Brazilian Diet (Phaseolus Vulgaris) According to Different Preparation Techniques.
Brief Title: Bioavailability of Proteins From Plant Based Diets
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eduardo Ferriolli (Other)
Responsible Party: Sponsor-Investigator, Eduardo Ferriolli, Assistant professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 2207
Record Dates: First submitted 2018-02-23; First posted 2018-04-10 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Protein Malabsorption; Nutrition Disorders; Sarcopenia
Keywords: protein availability; beans; children; elderly
MeSH Terms: conditions — Nutrition Disorders; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adults: Select the individual:
  Healthy, non-pregnant adults 18-65 years of age, not taking any medication, including NSAIDs, not taking antibiotics within 4 weeks of study, BMI within 18-35 range and stable weight.
  Exclusion criteria: children and elderly (over 65), pregnancy, diagnosed with non-communicable or communicable disease, being under restrictive diet, antibiotics within 4 weeks of study, medications within 4 weeks of study. They will eat beans for 5 days. The beans will be soaked for 3 h, water discarded and beans cooked for 20 min in pressure cook. And in the end for the week, adults will be eat the bean enrichment of deuterium for availability protein, collected urine, saliva and blood.
- Children: Fifty children will be recruited from ages varying from 1 to 3 years and of both sexes. Children who use medications, who do not habitually consume beans, will be excluded and when there is no explicit written authorization from the parents or guardians.
  All the children with different status of nutrition will be eaten the beans. They will eat beans for 5 days. The beans will be soaked for 3 h, water discarded and beans cooked for 20 min in pressure cook. And in the end for the week, children will be eat the bean enrichment of deuterium for availability protein, collected urine or saliva depend on the best biological samples of pilot study (adult).
- Elderly: Fifty individuals of both sexes will be recruited, previously evaluated by complete clinical / laboratory examination and medical history. The elderly will be excluded from antiinflammatory, chemotherapeutic, corticoid, allergy and bean aversion or antibiotic therapy. These drugs could interfere with protein bioavailability. They will eat beans for 5 days. The beans will be soaked for 3 h, water discarded and beans cooked for 20 min in pressure cook. And in the end for the week, elderly will be eat the bean enrichment of deuterium for availability protein, collected urine or saliva depend on the best biological samples of pilot study (adult).

SUMMARY:
The quality of protein intake has an important role within the nutritional needs of people throughout their lives around the world, particularly in developing countries and in particular during pregnancy and early childhood. It is likely that adequate protein reduce by 40% the prevalence of stunting (low height for age) in children under five years, according to World Health Organization data. Uncertainty about the quality of the diet, specifically with reference to quality proteins has potential impacts on health, economy, agriculture, and food security of a nation. The amino acid digestibility estimates based on stool analysis do not represent the amount of absorbed amino acid. Ideally, the bioavailable amino acid should be measured by methods that assess the difference between consumed and absorbed amino acids. However, the uptake of amino acids is not readily non-invasively measured in healthy humans. The use of vegetable protein intrinsically labeled by stable isotopes offers a solution to this problem. The deuterated water (2H2O), with relatively low cost, is suitable for labeling plant proteins such as those of beans. The labeled amino acids are present in the test meal ingested and incorporated into the blood, representing a single measure of bioavailability. This study aims to develop and apply a new methodology, using stable isotopes, to evaluate the bioavailability of bean protein, a very important food in the Brazilian diet, according to cooking procedures, through the use of deuterium. The project will be divided into two parts: a human nutrition and an agriculture part, the latter by planting/harvesting deuterium-labeled Phaseolus vulgaris L. After two weeks of blooming, deuterium water will be added to the bean crop, which will be subsequently dried. Chemical analysis and assessment of incorporation of deuterium in the beans will be done. Concurrent with the cultivation of beans, there will be a protein absorption test with 15 healthy volunteers for validation of the methods. For comparison purposes, milk protein labeled with deuterium and C13 will be used. The volunteers will consume the test meals. Blood, urine and saliva samples will be collected at baseline (before food ingestion), and in different times after the meal. In the next phase of this research, labeled beans produced by the agriculture experiment will be used to measure the protein absorption of volunteers of different groups (older persons, and stunting and non-stunting children). The samples will analyzed by isotope-ratio mass spectrometry. This methodology may promote a better understanding of the absorption of proteins and amino acids using less invasive methods in different age groups and clinical conditions. This work will have an important impact for the general population as well as for agriculture and health-related professionals.

DETAILED DESCRIPTION:
This study is divided in 4 phase. First Phase: Agriculture (Year 1) Site description: The experiment will carried out at the Experimental Farm of São Paulo's Agency for Agribusiness Technology (APTA) in Ribeirao Preto, Brazil, at the geographic coordinates of 21°12'26" S e 47°51'48" N and average altitude of 646 m. The annual rainfall is about 1427 mm, with average maximum and minimum temperature of 25°C and 19.3°C, respectively. The soil is classified as Oxitol with glay texture. The bean crop (Phaseolus vulgaris), will be grown at the 0,50m between rows with 12 seed per linear meters and at the 2 weeks after anthesis (flowering) the water supply will be amended with deuterium oxide to experimental development. The grain produced will be harvested to experimental analysis and consumption. The experimental area will have 5.000 m2 with common bean crop to produce enough quantity of grains to the experiment running. Seeds will be dried in a scale of 1 to 10 kg of dry and selected seeds.

Nutrients Composition Analysis (Year 1) Six samples of 100g each will be separated for nutrients composition analyses, that will be performed at the Animal Nutrition Laboratory of the Animal Science Institute of the University of São Paulo, Brazil. Right after harvesting, the food samples will be weighted and dried in a stove with forced air circulation at 65 degrees Celsius, during 72 hours. After this, samples will be ground in a mill with 2 mm hole sieve, and a subsample will be taken for the analysis of dry mass, protein, ether extract, mineral mass, energy, calcium and phosphorus, according to Official Methods of Analysis (AOAC) (1996). Fibre will be analysed in neutral and acid detergent according to reference Silva and Queiroz, 2005, and selenium will be analysed according to Olson et al., 1975. Energy analysis will be performed by a calorimetric bomb and fat by the extraction according to reference Bligh and Dyer, 1959, at the Nutrients Composition Laboratory of the Ribeirão Preto Medical School.

Second phase (pilot study), Nutrition Institute (Year 2) Subjects Fifteen adult volunteers will be recruited for method validation. Inclusion criteria

* Healthy, non-pregnant adults 18-65 years of age
* Not taking any medication, including NSAIDs
* Not taking antibiotics within 4 weeks of study
* BMI within 18-35 range
* Stable weight Exclusion criteria
* Children and elderly (over 65)
* Pregnancy
* Diagnosed with non-communicable or communicable disease
* Being under restrictive diet
* Antibiotics within 4 weeks of study
* Medications within 4 weeks of study Study design After approval of project by local ethics committee and obtaining signed informed consent, volunteers will be offered a test meal with milk protein. The test protein in the first place will be whole milk protein, produced with a low level deuterium enrichment within the study. This will permit the Carbon-13 single cell protein to be characterised against a well-studied animal protein known to possess high digestibility. Tracer Amino Acid (AA) appearance in the circulation (blood; saliva, urine and breath will also be sampled) and the relative appearance of test and reference protein will be taken as a measure of relative bioavailability which can be converted into an absolute measure once the reference protein has been characterised. The basic measurement will be of stable isotope enrichment in individual amino acids.

Phase 1 pilot study, Nutrition Institute. Fifteen adult volunteers will be recruited for method validation.

Third Phase is in 15 children (1-3 years, with different nutritional status) and Fourth phase is in 15 elderly (more than 65 years, with sarcopenia or not sarcopenia).

Test meal 1: Beans soaked for 3 h, water discarded and beans cooked for 20 min in pressure cook.

The test meal will be separated by the use for two weeks of unlabelled beans. The same approach as used in the pilot study of milk protein will be adopted to study the bioavailability of grain legumes through simultaneous comparison with a modest quantity carbon-13 enriched single cell protein combined in the same test meal.

All groups will be analysed food intake assessment, total urinary nitrogen and enrichment of deuterium in protein. Four 24h Recall Questionnaires will be applied to each volunteer during the periods of intake of the test meal, in order to verify the protein and calories consumption. Volunteers will be asked to keep their usual intake, to avoid changes in food consumption. Total urinary nitrogen of the samples will be analysed by the Kjeldahl method with ammonium micro diffusion. Compound specific isotope enrichment in amino acids will be analysed in saliva, urine, breath and blood samples. Carbon-13 in breath carbon dioxide (CO2) and Deuterium in urine enrichment will be analysed in Mass Spectrometry of Medicine School of Ribeirão Preto (FMRP-USP), Brazil, SP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-pregnant adults 18-65 years of age

  * Not taking any medication, including NSAIDs
  * Not taking antibiotics within 4 weeks of study
  * BMI within 18-35 range
  * Stable weight

Exclusion Criteria:

* Children and elderly (over 65)

  * Pregnancy
  * Diagnosed with non-communicable or communicable disease
  * Being under restrictive diet
  * Antibiotics within 4 weeks of study
  * Medications within 4 weeks of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Select healthy person with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-08-23 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Bioavailability protein using deuterium | It will be collected for 1 day
  Il will be measured new stable isotope method using deuterium for the study of the bioavailability of protein derived from beans in healthy adults, children and elderly. It will be assessed 45 persons, express in delta enrichment and analysis in Mass Spectrometry

SECONDARY OUTCOMES:
Bioavailability protein using carbon 13 | It will be collected for 1 day
  Il will be measured stable isotope using Carbon 13 for the study of the bioavailability of protein derived from beans in healthy adults, children and elderly. It will be assessed 45 persons, express in delta enrichment and analysis in Mass Spectrometry
Nutritional composition | through study completion in 1 week
  3 samples for beans cooked will be collected and will be verified the nutrients composition properties of the usually consumed Brazilian bean (Phaseolus vulgaris) labelled with deuterium like macronutrients and micronutrients in grams.

OTHER OUTCOMES:
Total urinary nitrogen | It will be collected for 1 day
  Urinary nitrogen of the samples will be analysed by the Kjeldahl method with ammonium micro diffusion

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ferriolli, PhD, Principal Investigator — São Paulo University, School of Medicine

IPD SHARING:
Plan to Share IPD: No
There is no plan to make this data available to other researchers. We will publish this data in the scientific magazine

REFERENCES:
- [Background] Elango R, Levesque C, Ball RO, Pencharz PB. Available versus digestible amino acids - new stable isotope methods. Br J Nutr. 2012 Aug;108 Suppl 2:S306-14. doi: 10.1017/S0007114512002498. PMID 23107543
- [Background] Hoffman DJ, Roberts SB, Verreschi I, Martins PA, de Nascimento C, Tucker KL, Sawaya AL. Regulation of energy intake may be impaired in nutritionally stunted children from the shantytowns of Sao Paulo, Brazil. J Nutr. 2000 Sep;130(9):2265-70. doi: 10.1093/jn/130.9.2265. PMID 10958822
- [Background] Gilani GS. Background on international activities on protein quality assessment of foods. Br J Nutr. 2012 Aug;108 Suppl 2:S168-82. doi: 10.1017/S0007114512002383. PMID 23107528